CLINICAL TRIAL: NCT03840525
Title: A Mind Body Intervention to Reduce Symptoms Among People Aging With HIV
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1R34AT009966-01 (NIH)
Record Dates: First submitted 2018-07-16; First posted 2019-02-15 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Mental Health; Physical Health
Keywords: qigong; HIV
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: The study will implement a 3 arm study including the qigong intervention, sham qigong intervention, and a treatment as usual condition. The qigong and sham qigong groups will be delivered virtually due to the coronavirus pandemic.
Who Masked: Participant
Masking Description: There will be a sham qigong arm of the study to mask qigong participation for the participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Qigong Intervention (Experimental): The qigong intervention consists of 1 hour/week qigong classes for 12 weeks to be delivered virtually. The first 2 weeks will include 2 hours/week classes. In addition, each participant will be instructed to practice qigong at home for 90 minutes.
  Interventions: Behavioral: The Qigong Intervention
- Sham Qigong (Sham Comparator): This group will also have 1 hour/weekly class delivered virtually that includes movements that are similar to qigong but will not include the meditation or breathwork that will be included in the actual qigong intervention arm.
  Interventions: Behavioral: Sham Qigong
- Treatment-as-usual (No Intervention): This group will receive no classes.

INTERVENTIONS:
Behavioral: The Qigong Intervention — Qigong is a low-impact, slow-movement, meditative form of exercise that has helped relieve mental and physical stressors.
  Arms: Qigong Intervention
Behavioral: Sham Qigong — This intervention includes similar body movements to qigong; however, it does not have the meditative or breath work.
  Arms: Sham Qigong

SUMMARY:
This study will develop and pilot test a qigong intervention with older people (50 and over) living with HIV. Participants (n=48) will be randomly assigned to one of 3 conditions: the qigong intervention, a sham qigong intervention, and a usual standard of care group. The study will determine the acceptability and feasibility of the study. If found effective, the qigong intervention will also improve the psychological and physical symptoms of older people living with HIV.

DETAILED DESCRIPTION:
Half of those infected with HIV in the United States are over 50 years of age; this is expected to increase to 70% by 2020. Yet, few interventions exist for older people living with HIV/AIDS that address psychological symptoms, and none that address physical symptoms, both of which are prevalent in this population. There is a need to find innovative and accessible interventions that can help older people living with HIV/AIDS to manage their symptoms. Mind-body interventions, like Tai chi and Qi gong (TCQ), improves both physical and psychological health, and might also promote immune functioning. TCQ is a series of slow, low-impact meditative movements that integrates breath work, meditation, and stances. The investigators propose the refinement, adaptation, acceptability and feasibility testing of a standardized TCQ intervention shown efficacious with cancer patients, to an ethnically diverse population of older people living with HIV/AIDS, with the goal of enhancing their ability to manage psychological and physical symptoms. Thus, this study proposes three aims: (i) to refine and culturally adapt a TCQ intervention protocol for a diverse sample of older people living with HIV/AIDS (50 years of age or older); (ii) to evaluate the acceptability and feasibility of the TCQ intervention, a sham qigong control condition, and a standard of care control condition for older people living with HIV/AIDS (n = 48); and (iii) explore any preliminary evidence of efficacy of the TCQ intervention and the control conditions on alleviating physical and psychological symptoms. Participants will be recruited from a federally qualified health center in Miami, Florida. Adaptation of the TCQ intervention, the first aim, will be done through qualitative research. An expert panel discussion, key informant interviews, and three focus groups will be conducted, and analyzed by thematically based content analysis. To address aims 2 and 3, the investigators will conduct a pilot study; participants will be randomized to one of 3 conditions: the TCQ intervention, a sham qigong condition, and a standard of care condition. This is a pilot study to assess feasibility, acceptability, and preliminary efficacy, therefore, analyses will be primarily descriptive. The investigators will assess feasibility and acceptability through questionnaires and adherence to TCQ. The investigators will assess preliminary evidence of efficacy by looking at instruments that measure depression, anxiety, social support, as well as clinical outcomes. These will be described through proportions, means, and changes over time through graphing techniques. Outcomes will be assessed at baseline, post-intervention, and at three months follow up. The investigators will conduct preliminary models that will provide information on estimating effect size and power needed for a larger clinical trial. Note: Due to the coronavirus pandemic, this intervention was adapted from an in-person intervention to a virtual intervention. The intervention is exactly the same except for the difference in delivery method.

ELIGIBILITY:
Inclusion Criteria:

* 50 year or older;
* HIV+,
* able to provide consent;
* must have reliable internet access; and
* willing to participate for the length of the intervention.

Exclusion criteria.

* Participants who are unable to stand for 10-minute segments (i.e., wheelchair or walker bound); and
* participants who have substantial (regular weekly practice for more than 3 months in the past 12 months) experience with mind-body interventions will be excluded because the control group may be contaminated by prior experience.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Borinquen Medical Centers of Miami Dade, Miami, Florida, United States

REFERENCES:
- [Derived] Ibanez GE, Fennie K, Larkey L, Hu N, Algarin AB, Valdivia C, Lavretsky H. A tai chi/qigong intervention for older adults living with HIV: a study protocol of an exploratory clinical trial. Trials. 2020 Sep 22;21(1):804. doi: 10.1186/s13063-020-04728-x. PMID 32962749

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Qigong Intervention | Sham Qigong | Treatment-as-usual
Started | 16 | 16 | 16
Completed | 13 | 12 | 10
Not Completed | 3 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Qigong Intervention | Sham Qigong | Treatment-as-usual | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (6.0) | 61.0 (6.0) | 61.0 (4.0) | 60.0 (5.0)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The baseline data for 1 participant (assigned to the sham control group) was lost by accident.
  Participants
    Gender: number analyzed (Participants) | 16 | 15 | 16 | 47
    Gender: Male | 8 | 9 | 9 | 26
    Gender: Female | 6 | 6 | 7 | 19
    Gender: Transgender/Other | 2 | 0 | 0 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The baseline data for 1 participant (assigned to the sham control group) was lost by accident.
  Participants
    Race: number analyzed (Participants) | 16 | 15 | 16 | 47
    Race: White | 9 | 7 | 8 | 24
    Race: Black | 7 | 8 | 8 | 23
Region of Enrollment [Number; unit: participants] — Population: The baseline data for 1 participant (assigned to the sham control group) was lost by accident.
  participants
    United States: number analyzed (Participants) | 16 | 15 | 16 | 47
    United States | 16 | 15 | 16 | 47

OUTCOME MEASURES:

1. Primary Outcome: Acceptability: Satisfaction With Weekly Intervention Sessions
Description: Satisfaction were measured by asking the following questions after each session: "I really enjoyed today's class"; "Today's class met my expectations"; "The instructor was engaged in today's class". Responses are on a 5 point Likert scale (1=strongly disagree to 5=strongly agree) with lower scores meaning less satisfaction. Both the qigong intervention and the sham qigong control group will be asked these satisfaction items. Acceptability was defined as responding either agree (4) or strongly agree (5) to each of these items. Therefore, participants who had an average score of at least 4.00 across all 12 weekly groups was considered a participant that found the intervention acceptable. The number of participants who found the intervention is counted below.
Time Frame: Assessments were conducted at Week 1 to Week 12 (i.e., once a week for 12 weeks). All weekly scores were averaged across weeks. The number of participants with an average score of 4.00 or higher found the intervention acceptable and is reported below
Population: The treatment as usual group is 0 because they did not receive any classes. Only the qigong intervention and the sham qigong groups were asked these items because they are the only ones receiving classes.
Measure: Count of Participants; unit: Participants
Arm/Group | Qigong Intervention | Sham Qigong | Treatment-as-usual
Number analyzed (Participants) | 13 | 13 | 0
Participants
  Acceptability: Enjoyed classes | 13 | 12 | 0
  Acceptability: Class met expectations | 12 | 13 | 0
  Acceptability: Instructor engaged | 13 | 12 | 0
Statistical Analysis 1: Comparison: Qigong Intervention vs Sham Qigong; Test type: Equivalence — To estimate precision, 95%CI will be calculated using Wilson's score method, which uses asymptotic variance and is appropriate for small sample sizes100. The formula is as follows: (2np + z2 ± √(z2 + 4npq)) / 2(n+ z2). If the proportion of participants who rate the intervention as acceptable is 80% or greater, we will consider the intervention acceptable; Descriptive statistics were conducted. No group comparisons were done due to the fact that this was a feasibility trial and not an efficacy trial. 80% was used as the benchmark for acceptability

2. Primary Outcome: Acceptability: Are Participants Doing Home Practice Sessions at 2 Week Post Intervention
Description: Acceptability was measured by asking the following question at 2 weeks post intervention (Week 14): Did you practice at home this week? Response format is yes=1, no=0 . This outcome determines if the participants continued their home practice of Qigong 2 weeks after the end of the intervention. The number of participants who responded yes were summed and reported below. The intervention was deemed acceptable to participants if at least 80% of participants were still practicing at home at Week 14.
Time Frame: Assessment was conducted 2 week post intervention (Week 14)
Population: The treatment as usual group is 0 because they did not receive any classes to practice. The sample size for the qigong and the sham qigong groups reflect the number of participants that completed the 2 week post intervention assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Qigong Intervention | Sham Qigong | Treatment-as-usual
Number analyzed (Participants) | 11 | 9 | 0
Participants | 8 | 6 | 0
Statistical Analysis 1: Comparison: Qigong Intervention vs Sham Qigong; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Descriptive statistics was conducted to determine acceptability for both the qigong and sham qigong group. No between group comparisons were conducted. A benchmark of 80% was used to determine acceptability

3. Primary Outcome: Acceptability: Session Attendance (Reported as Percentages)
Description: The investigators collected attendance after each weekly session (Week 1 to Week 12). An average attendance across all weekly sessions was calculated by taking the number of groups attended divided by the number of total sessions possible. The intervention was deemed acceptable if participants attended at least 70% of the weekly groups. The number of participants who attended 70% of the weekly groups were summed and reported below.
Time Frame: Assessments were conducted at Week 1 up to Week 12 (i.e., once a week after each session).
Population: The treatment as usual group was not analyzed since they did not receive any classes and therefore had no attendance.
Measure: Count of Participants; unit: Participants
Arm/Group | Qigong Intervention | Sham Qigong | Treatment-as-usual
Number analyzed (Participants) | 16 | 16 | 0
Participants | 10 | 9 | 0
Statistical Analysis 1: Comparison: Qigong Intervention vs Sham Qigong; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Descriptive statistics were conducted to determine acceptability. Benchmark for acceptability was set at 80% of participant attending at least 70% of the classes

4. Primary Outcome: Frequency of Home Practice Sessions at 2 Weeks Post Intervention (Week 14)
Description: The investigators collected information on how often participants practiced at home at two weeks post intervention (Week 14). At Week 14, participants were asked 'If you are practicing at home, how often did you practice the movements?' Response format is: 1=very frequent (every day), 2=frequent (a few times a week), 3=infrequent (once a week), and 4=very infrequent (less than once a week). Scores were averaged with the acceptability benchmark being that participants who practiced very frequently (1) or frequently (2) found the intervention acceptable. That is, participants whose average score was 2.00 or less considered the intervention acceptable. The number of participants who found the intervention acceptable were summed and reported below.
Time Frame: Assessments were conducted once at 2 week post intervention (Week 14).
Population: Analysis population is based on participants who completed the 2 week follow up assessment and who reported practicing the movements.
Measure: Count of Participants; unit: Participants
Arm/Group | Qigong Intervention | Sham Qigong | Treatment-as-usual
Number analyzed (Participants) | 8 | 6 | 0
Participants | 6 | 4 |

5. Primary Outcome: Acceptability: Frequency of Home Practice Sessions at Week 24 (3 Months Post Intervention)
Description: The investigators collected information on how frequently the participants were practicing the intervention at home at Week 24. Participants were asked the following: "If practicing at home in the last 3 months, how often have you practiced the movements?" Responses were 1=very frequently (every day), 2= frequently (a few times a week), 3=infrequently (once a week), or 4=very infrequently (less than once a week). Acceptability was determined if at least 70% of the participants reported very frequently (1) or frequently (2) home practice at Week 24. Participants with scores of 2.00 or less on this item were summed and then divided by the number of participants who reported any home practice in the last 3 months and also completed an assessment at Week 24.
Time Frame: Outcome was measured at Week 24 (i.e., 3 month post intervention)
Population: Participants in the Treatment as usual group was not analyzed because they did not receive any group sessions or instructions so there were no movements to practice at home.
Measure: Count of Participants; unit: Participants
Arm/Group | Qigong Intervention | Sham Qigong | Treatment-as-usual
Number analyzed (Participants) | 10 | 6 | 0
Participants | 7 | 5 | 0

6. Primary Outcome: Acceptability: Home Practice of the Intervention at Week 24 (3 Months Post Intervention)
Description: The investigators collected information on home practice sessions at Week 24 (the 3 month follow up assessment. Participants were asked the following: "have you practiced any of the movements in the last 3 months?" Response format was No=0, Yes=1. The acceptability benchmark was set at 70%. If at least 70% of participants reported any home practice at 3 months (Week 24) post intervention, the intervention would be deemed acceptable. The number of participants were summed and then divided by the number of participants assigned to the participant's study group assignment and who completed an assessment at week 24 in order to calculate a percentage.
Time Frame: Outcome was measured at Week 24 (3 month post intervention).
Population: The treatment as usual control group did not receive any group sessions so there was no home practice to report.
Measure: Count of Participants; unit: Participants
Arm/Group | Qigong Intervention | Sham Qigong | Treatment-as-usual
Number analyzed (Participants) | 13 | 13 | 0
Participants | 10 | 6 | 0

7. Secondary Outcome: Change in Mental Health at 2 Weeks Post Intervention
Description: Mental Health will be assessed using the following standardized scale: the Depression Anxiety & Stress Scale (Ng, et al.; DASS-21 items). The DASS responses range from 0-3. The total score ranges from 0-42, with higher scores reflecting more severe symptoms
Time Frame: Assessments will be conducted at baseline, 2 weeks post intervention
Reporting Status: Not Posted

8. Secondary Outcome: Change in Mental Health at 3 Months Post Intervention
Description: as for outcome 7
Time Frame: Assessments will be conducted at baseline, 3 months post intervention
Reporting Status: Not Posted

9. Secondary Outcome: Change in Physical Health Status as Measured by The Revised Sign & Symptom Check-List for HIV (Holzemer, et al.; 45 Items) at 2 Weeks Post Intervention
Description: Physical Health will be assessed using the following standardized scale: The Revised Sign & Symptom Check-List for HIV (Holzemer, et al.; 45 items). The Symptoms Checklist total scores range from 0-135, with greater scores reflecting more symptoms.
Time Frame: Assessments will be conducted at baseline, 2 weeks post intervention
Reporting Status: Not Posted

10. Secondary Outcome: Change in Physical Health Status as Measured by The Revised Sign & Symptom Check-List for HIV (Holzemer, et al.; 45 Items) at 3 Months Post Intervention
Description: as for outcome 9
Time Frame: Assessments will be conducted at baseline, 3 months post intervention
Reporting Status: Not Posted

11. Secondary Outcome: Change in Physical Health Status as Measured by The HIV-related Fatigue Scale (Belza, et al.,16 Items) at 2 Weeks Post Intervention
Description: Physical Health will be assessed using the following standardized scale: The HIV-related Fatigue Scale (Belza, et al.,16 items) . The total score for the Fatigue Scale ranges from 0-50, with greater scores reflecting more fatigue.
Time Frame: Assessments will be conducted at baseline, 2 weeks post intervention
Reporting Status: Not Posted

12. Secondary Outcome: Change in Physical Health Status as Measured by The HIV-related Fatigue Scale (Belza, et al.,16 Items) at 3 Months Post Intervention
Description: as for outcome 11
Time Frame: Assessments will be conducted at baseline, 3 months post intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the duration of the clinical trials: from enrollment (baseline interview) through the intervention phase (3 months), and until study completion (3 month post intervention). Therefore, adverse event data were collected for 6 months.
Arm/Group | Qigong Intervention | Sham Qigong | Treatment-as-usual
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/16 | 1/16
Other Adverse Events (participants affected / at risk) | 1/16 | 0/16 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Qigong Intervention (N=16) | Sham Qigong (N=16) | Treatment-as-usual (N=16)
Hospitalization (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) — Participant was briefly hospitalized. Reasons for hospitalization was related to their HIV status. This event was not study-related.
Kidney biopsy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) — Participant reported an outpatient medical procedure, specifically a kidney biopsy. This event was not deemed study-related.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Qigong Intervention (N=16) | Sham Qigong (N=16) | Treatment-as-usual (N=16)
Participant experience soreness due to intervention (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) — Participant reported feeling severe soreness from the physical activity in the TCQ intervention. This event was deemed study-related; however, the participant only reported soreness twice and was able to continue the study and complete the study.

LIMITATIONS AND CAVEATS:
Sample size was reduced, with NIH approval, due to the Covid-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03840525/Prot_SAP_000.pdf